CLINICAL TRIAL: NCT02458625
Title: A Comparison Between Intravenous Iron Sucrose to Its Combination With Oral Iron Supplements for the Treatment of Postpartum Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Zohar Nachum, MD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0133-14
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Postpartum Anemia
MeSH Terms: interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron sucrose 500 mg (Active Comparator): One treatment arm will receive a single dose of I.V iron sucrose 500 mg.
  Interventions: Dietary Supplement: Iron sucrose 500 mg
- Iron sucrose 500 mg+60 mg Iron bisglycinate (Active Comparator): Second treatment arm will receive a single dose of I.V iron sucrose 500 mg and oral treatment with 60 mg Iron bisglycinate for 6 weeks after giving birth.
  Interventions: Dietary Supplement: Iron sucrose 500 mg; Dietary Supplement: Iron bisglycinate 60 mg

INTERVENTIONS:
Dietary Supplement: Iron sucrose 500 mg
Dietary Supplement: Iron bisglycinate 60 mg
  Arms: Iron sucrose 500 mg+60 mg Iron bisglycinate

SUMMARY:
This study is aimed to compare the efficacy of two mode of iron administration to treat post partum anemia - a single dose of intravenous iron sucrose versus a single dose of iron sucrose and 6 weeks of treatment with oral iron supplement.

DETAILED DESCRIPTION:
Anemia is common following delivery. It is associated with disturbing symptoms such as fatigue, cognitive impairment and syncope in severe cases. International guidelines recommend to use intravenous iron sucrose to treat intermediate and severe anemia until the target hemoglobin is achieved. However, patient's compliance after delivery is low, making the administration of several doses difficult. In those cases oral iron supplements might be used. In the present study the investigators will compare the efficacy of two iron administration protocols to treat post partum anemia - a single dose of intravenous iron sucrose versus a single dose of iron sucrose and 6 weeks of treatment with oral iron supplement.

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 years old after giving birth
* Women who suffer from iron deficiency anemia, defined as hemoglobin< 9.5 g/dl without one of the conditions that are described in the exclusion criteria

Exclusion Criteria:

* Women who suffer from known allergy for iron supplements
* Women who suffer from anemia not due to iron deficiency
* Women who suffer from acute infection
* Women who suffer from liver failure or viral hepatitis
* Women who suffer from thalassemia or hemoglobinopathies
* Women who suffer from renal failure
* Women who suffer from unbalanced thyroid disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
The change between the hemoglobin level at randomization and the hemoglobin level after 6 weeks postpartum | After 6 weeks post partum

SECONDARY OUTCOMES:
Women's satisfaction from the protocol treatment according to the VAS (visual analog scale) after 6 weeks post partum | Up to 6 weeks post partum
The composite symptoms of anemia and functional capacity after 6 weeks postpartum as assessed by a questionnaire | six weeks post partum
Type and rate of adverse events | Up to 6 weeks post partum
The rate of patients who discontinued treatment | Up to 6 weeks post partum
The change in hemoglobin level, ferritin, serum iron, transferrin, MCV and iron saturation from randomization to 6 weeks post partum | From randomization to 6 weeks post partum
The rate of women who will reach a target hemoglobin of at least 12 g/dl after 6 weeks of treatment | Six weeks post partum

CONTACTS AND LOCATIONS:
Locations (1):
- Emek Medical Center, Afula, Israel

REFERENCES:
- [Derived] Yefet E, Mruat Rabah S, Sela ND, Hosary Mhamed S, Yossef A, Nachum Z. Addition of oral iron bisglycinate to intravenous iron sucrose for the treatment of postpartum anemia-randomized controlled trial. Am J Obstet Gynecol. 2021 Dec;225(6):668.e1-668.e9. doi: 10.1016/j.ajog.2021.06.069. Epub 2021 Jun 23. PMID 34171389